CLINICAL TRIAL: NCT05367492
Title: Randomized Controlled Trial of Varenicline for Cessation of Nicotine Vaping in Adolescent Non-smokers
Brief Title: Varenicline for Nicotine Vaping Cessation in Adolescents
Acronym: ViVA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Anne Eden Evins, Founder Director, Center for Addiction Medicine and Director for Faculty Development, Department of Psychiatry; Cox Family Professor of Psychiatry in the Field of Addiction Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020P002774; R01DA052583 (NIH)
Record Dates: First submitted 2022-05-04; First posted 2022-05-10 (Actual); Results first posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Vaping; Nicotine Dependence
Keywords: Vaping; Nicotine; Adolescents; Cessation; Varenicline
MeSH Terms: conditions — Vaping; Tobacco Use Disorder

STUDY DESIGN:
Intervention Model Description: Up to 300 participants will be consented and approximately 225 participants will be randomized in a double blind, placebo-controlled, parallel-group trial comparing vaping abstinence rates in participants randomly assigned to (1) varenicline added to behavioral and texting support for vaping cessation (V+BC) and (2) identical placebo added to behavioral and texting support for vaping cessation (P+BC) (primary comparison). Exploratory secondary comparisons will be made between double blind arms 1 and 2 and the single blind (3) enhanced usual care arm.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Eligible participants will be assigned to one of three groups using a computer-generated randomization code conducted by MGH Research Pharmacy personnel with no other interactions with participants.
  The full randomization code of the two double blind treatment arms (arm 1 active varenicline and arm 2 identical placebo), and the single blind EUC arm (arm 3) will be held in the MGH research pharmacy and available to study PIs for urgent medical need only. Participants, investigators and outcome assessors will be fully blind to all 3 arms.
  A partial randomization code identifying those assigned to double-blind treatment (a combined list of study IDs assigned to either study arm 1 or 2) vs single blind EUC (study arm 3) will be held by a scheduler who is not associated with outcomes assessment, data analysis or interpretation. Assignment to Arm 3, single blind EUC only, will be masked to investigators and outcomes assessors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Double Blind Varenicline (V + BC) (Experimental): Participants will...
  * Receive the drug varenicline, in tablet form, up to 1 mg BID for 12 weeks.
  * Attend QuitVaping behavioral support sessions, completed in-person or via video-conferencing, once per week for 12 weeks.
  * Be encouraged to sign up for This Is Quitting (TIQ), a text message vaping cessation program for adolescents.
  Interventions: Drug: Double Blind Varenicline; Behavioral: QuitVaping; Behavioral: This Is Quitting
- Double Blind Placebo (P + BC) (Placebo Comparator): Participants will...
  * Receive placebo tablets, identical in appearance to varenicline, up to 1 mg BID for 12 weeks.
  * Attend QuitVaping behavioral support sessions, completed in-person or via video-conferencing, once per week for 12 weeks.
  * Be encouraged to sign up for This Is Quitting (TIQ), a text message vaping cessation program for adolescents.
  Interventions: Drug: Double Blind Placebo; Behavioral: QuitVaping; Behavioral: This Is Quitting
- Single Blind Enhanced Usual Care (EUC) (Active Comparator): Participants will...
  * Receive NO drug intervention.
  * Attend NO behavioral support sessions.
  * Be encouraged to sign up for This Is Quitting (TIQ), a text message vaping cessation program for adolescents.
  Interventions: Behavioral: This Is Quitting

INTERVENTIONS:
Drug: Double Blind Varenicline — For participants 16-17 years old, ≤ 55 kg:
  * 0.5 mg once daily for 7 days, then
  * 0.5 mg twice daily for 11 weeks
  For participants 16-17 years old, >55 kg:
  * 0.5 mg once daily or 3 days,
  * 0.5 mg twice daily for 4 days
  * 1.0 mg twice daily for 11 weeks
  For participants 18+ years old:
  * 0.5 mg once daily or 3 days,
  * 0.5 mg twice daily for 4 days
  * 1.0 mg twice daily for 11 weeks
  Arms: Double Blind Varenicline (V + BC)
Drug: Double Blind Placebo — For participants 16-17 years old, ≤ 55 kg:
  * 0.5 mg once daily for 7 days, then
  * 0.5 mg twice daily for 11 weeks
  For participants 16-17 years old, >55 kg:
  * 0.5 mg once daily or 3 days,
  * 0.5 mg twice daily for 4 days
  * 1.0 mg twice daily for 11 weeks
  For participants 18+ years old, regardless of weight:
  * 0.5 mg once daily or 3 days,
  * 0.5 mg twice daily for 4 days
  * 1.0 mg twice daily for 11 weeks
  Arms: Double Blind Placebo (P + BC)
Behavioral: QuitVaping — QuitVaping is a manualized intervention based on the American Lung Association smoking cessation program modified with adolescent appropriate content and language for vaping cessation from the vaping section of teen.smokefree.gov and the Truth Initiative. These behavioral support sessions will be delivered weekly during the 12-week treatment phase via videoconference or in- person.
  Arms: Double Blind Placebo (P + BC); Double Blind Varenicline (V + BC)
Behavioral: This Is Quitting — A free, publicly available text message vaping cessation program from Truth Initiative, designed specifically to help adolescents who vape nicotine quit. Participants who set a quit date receive messages for a week preceding it and 30 days afterward that include encouragement and support, skill- and self-efficacy building exercises, coping strategies, and information about the risks of vaping, benefits of quitting and cutting down to quit.
  Other Names: TIQ

SUMMARY:
The study will test the hypothesis that varenicline, when added to behavioral and texting support for vaping cessation, will improve vaping abstinence rates in adolescents dependent on vaped nicotine over placebo plus behavioral and texting support for vaping cessation. Approximately 225 adolescents will be randomly assigned to one of three arms (1) varenicline up to 1 mg bid for 12 weeks plus behavioral and texting support for vaping cessation (V+BC), (2) identical appearing placebo plus behavioral and texting support (P+BC) and (3) enhanced usual care (EUC). The primary comparison will be the double-blind, placebo-controlled comparison of vaping cessation rates in those assigned to varenicline vs placebo.

DETAILED DESCRIPTION:
Up to 300 adolescents, aged 16-25, who vape, do not smoke regularly, and want to quit vaping will be consented; approximately 225 eligible participants will be randomly assigned to a double blind, placebo-controlled intervention consisting of (1) varenicline or (2) identical placebo, up to 1 mg bid for 12 weeks, plus behavioral and texting support for adolescent vaping cessation or to (3) enhanced usual care. The primary comparison of interest is the double blind, placebo-controlled efficacy comparison of those assigned to (1) varenicline vs (2) placebo on vaping abstinence outcomes. The secondary comparison of placebo plus behavioral and texting support vs. EUC will estimate the efficacy of behavioral and texting support for vaping cessation in this population. The secondary comparison of varenicline plus behavioral and texting support vs EUC will estimate of the efficacy of varenicline treatment plus behavioral and texting support for vaping cessation in this population vs no treatment, the most common vaping cessation intervention. All participants will complete enrollment and baseline visits, and six monthly assessment visits. Those assigned to double blind intervention (study arms 1 or 2) will also complete 12 weekly behavioral support sessions. Assessors will be blind to intervention assignment (arm 1 or 2) vs EUC (arm 3) assignment. Among those assigned to the V+BC or P+BC intervention arms, study staff and participants will be blind to active varenicline vs placebo assignment, such that among those assigned to intervention (arm 1 or 2), assignment to study drug will be double blind. For those assigned a double blind intervention arm, study staff will distribute varenicline or identical appearing placebo and give instructions use at weeks 0, 2, 4 and 8. Participants will be asked to bring all empty and unused study medication at each in-person study visit through Week 12. The enrollment visit will consist of questionnaires, diagnostic assessments, vitals, saliva and urine samples. The baseline visit will consist of questionnaires, a saliva sample for cotinine concentration, and randomization. Monthly visits will consist of interviews, questionnaires and a saliva and urine sample. Weekly treatment meetings for participants assigned to arms 1 or 2 will consist of cognitive behavioral support and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Ages 16-25, inclusive;
* Self-report of daily or near daily nicotine vaping for the prior ≥ 3 months and semi-quantitative saliva screening for cotinine positive for recent nicotine use;
* Nicotine dependence as defined by a score ≥4 on the 10-item E-cigarette Dependence Inventory (ECDI), or report of persistent use despite negative consequences, or prior failed quit attempts;
* Self-report of no regular combusted tobacco use in the past 2 months at enrollment and exhaled CO <10 ppm;
* Total body weight at enrollment ≥35 kg (77 lbs);
* Report willingness to try varenicline to stop vaping;
* Able to understand study procedures and read and write in English;
* Have a parent or legal guardian who is able and willing to provide written informed consent (if under the age of 18);
* Competent and willing to provide written informed consent (if age 18+) or assent (if under 18);
* For participants who could become pregnant: negative urine pregnancy test at enrollment and agree to use effective contraception (e.g., abstinence, hormonal contraception, intra-uterine device, sterilization, or double barrier contraception) during the study.

Exclusion Criteria:

* Use of a smoking cessation medication in the prior month (nicotine patch, gum, nasal spray, or inhaler, varenicline, bupropion);
* Unwilling to abstain during the study from using smoking cessation aids other than those provided by the study;
* Unstable medical condition, epilepsy, severe renal impairment;
* Inpatient psychiatric hospitalization in the prior 6 months, serious suicidal ideation or suicide attempt within 6 months of enrollment, recent active suicidal ideation or suicidal behavior identified at enrollment or baseline visits;
* Evidence of active problem substance use severe enough to compromise ability to safely participate, in the investigator's opinion;
* Prior adverse drug reaction to varenicline;
* Unwilling to provide urine samples;
* Any condition or situation that would, in the investigator's opinion, make it unlikely that the participant could adhere safely to the study protocol;
* Ward of the state.

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 261 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eden Evins, MD, Principal Investigator — Massachusetts General Hospital; Randi Schuster, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Center for Addiction Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study are available upon request. Data will include de-identified individual patient-level data, a data dictionary, and analytic code. Investigators proposing to use the data must execute a data use agreement with Massachusetts General Hospital and have approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, before data is shared. Data will be available within three months of manuscript publication. Requests for data should be sent to aeevins@mgh.harvard.edu or rschuster@mgh.harvard.edu.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following manuscript publication.
Access Criteria: Researchers who provide a methodologically sound proposal to achieve aims in the approved proposal. Data use agreement and approval from an Institutional Review Board, Independent Ethics Committee, or Research Ethics Board are required.

REFERENCES:
- [Background] Schuster RM, Cather C, Pachas GN, Nielsen L, Iroegbulem V, Dufour J, Potter K, Levy S, Gray KM, Evins AE. A randomized controlled trial of varenicline and brief behavioral counseling delivered by lay counselors for adolescent vaping cessation: Study protocol. Front Psychiatry. 2023 Mar 15;14:1083791. doi: 10.3389/fpsyt.2023.1083791. eCollection 2023. PMID 37009114
- [Derived] Gilman JM, Cather C, Reeder HT, Evohr B, Pachas GN, Gray KM, McClure EA, Schuster RM, Evins AE. Cannabis Use and Nicotine Vaping Cessation Outcomes: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2025 Dec 1;8(12):e2547799. doi: 10.1001/jamanetworkopen.2025.47799. PMID 41385228
- [Derived] Evins AE, Cather C, Reeder HT, Evohr B, Potter K, Pachas GN, Gray KM, Levy S, Rigotti NA, Iroegbulem V, Dufour J, Casottana K, Costello MA, Gilman JM, Schuster RM. Varenicline for Youth Nicotine Vaping Cessation: A Randomized Clinical Trial. JAMA. 2025 Jun 3;333(21):1876-1886. doi: 10.1001/jama.2025.3810. PMID 40266580

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial recruited participants from a single U.S. state from June 2022 to November 2023.
Groups:
- Double Blind Varenicline (V+BC): Participants will...
  * Receive the drug varenicline, in tablet form, up to 1 mg BID for 12 weeks.
  * Attend QuitVaping behavioral support sessions, completed in-person or via video-conferencing, once per week for 12 weeks.
  * Be encouraged to sign up for This Is Quitting (TIQ), a text message vaping cessation program for adolescents.
- Double Blind Placebo (P+BC): Participants will...
  * Receive placebo tablets, identical in appearance to varenicline, up to 1 mg BID for 12 weeks.
  * Attend QuitVaping behavioral support sessions, completed in-person or via video-conferencing, once per week for 12 weeks.
  * Be encouraged to sign up for This Is Quitting (TIQ), a text message vaping cessation program for adolescents.
Period: Study Intervention (Week 12)
Arm/Group | Double Blind Varenicline (V+BC) | Double Blind Placebo (P+BC) | Single Blind Enhanced Usual Care (EUC)
Started | 88 | 87 | 86
Completed | 88 | 83 | 85
Not Completed | 0 | 4 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 2 | 1
Period: Study Follow Up (Week 24)
Arm/Group | Double Blind Varenicline (V+BC) | Double Blind Placebo (P+BC) | Single Blind Enhanced Usual Care (EUC)
Started | 88 | 83 | 85
Completed | 88 | 81 | 85
Not Completed | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Double Blind Varenicline (V+BC) | Double Blind Placebo (P+BC) | Single Blind Enhanced Usual Care (EUC) | Total
Number analyzed (Participants) | 88 | 87 | 86 | 261
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.6 (2.0) | 21.4 (2.1) | 21.4 (2.0) | 21.5 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 47 | 46 | 139
  Male | 42 | 40 | 40 | 122
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 18 | 8 | 43
  Not Hispanic or Latino | 71 | 69 | 78 | 218
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 13 | 17 | 18 | 48
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 7 | 4 | 16
  White | 56 | 49 | 55 | 160
  More than one race | 10 | 10 | 8 | 28
  Unknown or Not Reported | 4 | 3 | 1 | 8
Region of Enrollment [Number; unit: participants]
  United States | 88 | 87 | 86 | 261
Post-secondary School [Count of Participants; unit: Participants] | 86 | 85 | 86 | 257
E-cigarette use: Median number of days used per week in last 30 days [Median (Inter-Quartile Range); unit: days per week] — The median number of days per week in which a participant used e-cigarettes in last 30 days. E-cigarette use (frequency, amount) was assessed using timeline followback methods. Population: Due to technical issues with the timeline followback application, data was lost for 7 participants.
  days per week
    number analyzed (Participants) | 87 | 84 | 83 | 254
    (all) | 7 [7 to 7] | 7 [7 to 7] | 7 [7 to 7] | 7 [7 to 7]
E-Cigarette Dependence Inventory (ECDI) [Mean (Standard Deviation); unit: total score on a scale] — The Penn State Electronic Cigarette Dependence Inventory (ECDI) is a 10-item validated measure assessing electronic cigarette dependency. Scores range from 0 to 20. Higher scores indicate greater dependence. Scores indicate the following: Not dependent [score 0-3], low dependence [score 4-8], medium dependence [score 9-12], and high dependence [score ≥13].
  total score on a scale | 12.5 (3.8) | 13.7 (4.0) | 12.8 (3.8) | 13.0 (3.9)
Motivation to Quit Vaping [Mean (Standard Deviation); unit: score on a scale] — Motivation to quit vaping was assessed by a single-item scale from the PhenX Toolkit with scores of 1 to 10. The item reads "How motivated are you to quit vaping on a scale where 1= not at all motivated and 10= extremely motivated". Higher scores indicate greater motivation to quit.
  score on a scale | 7.1 (1.7) | 6.7 (1.8) | 7.1 (1.6) | 7.0 (1.7)
Minnesota Nicotine Withdrawal Scale (MNWS) [Mean (Standard Deviation); unit: score on a scale] — The Minnesota Nicotine Withdrawal Scale (MNWS) is an 8-item measure assessing the severity of nicotine withdrawal symptoms. Items are scored on an ordinal scale from 0 ("not at all") to 4 ("extreme") with total scores ranging from 0 to 32. Higher scores indicate greater severity of nicotine withdrawal symptoms.
  score on a scale | 10.5 (6.1) | 10.6 (6.1) | 11.2 (6.0) | 10.8 (6.0)
Questionnaire of Vaping Craving (QVC) [Mean (Standard Deviation); unit: score on a scale] — The Questionnaire of Vaping Craving is a 10-item measure used to assess desire and intent to vape and anticipation of positive outcomes from vaping. Each item is scored on a 7-point Likert scale from 1 ("strongly disagree") to 7 ("strongly agree") with total scores ranging from 10 to 70. Higher scores indicate greater vaping craving.
  score on a scale | 41.3 (11.5) | 42.3 (13.1) | 38.5 (13.8) | 40.7 (12.9)
Combusted Tobacco: Past 30-day use [Count of Participants; unit: Participants] — Count of participants who reported using any combusted tobacco in the past 30 days. Past 30-day combusted tobacco use was assessed using timeline followback methods. Population: Due to technical issues with the timeline followback application, data was lost for 5 participants.
  Participants
    number analyzed (Participants) | 86 | 87 | 83 | 256
    (all) | 6 | 7 | 8 | 21
Combusted Tobacco: Median number of days used per week in last 30 days [Median (Inter-Quartile Range); unit: days per week] — The median number of days per week in which a participant used combusted tobacco in the last 30 days. Combusted tobacco use (frequency, amount, type) was assessed using timeline followback methods. Population: Due to technical issues with the timeline followback application, data was lost for 7 participants.
  days per week
    number analyzed (Participants) | 85 | 86 | 83 | 254
    (all) | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
Lifetime cigarettes smoked ≥100 [Count of Participants; unit: Participants] — Count of participants who report smoking 100 or more cigarettes in their lifetime. Lifetime cigarette use was assessed by self-report measure.
  Participants | 9 | 7 | 5 | 21
Cannabis: Past 30-day use [Count of Participants; unit: Participants] — Count of participants reporting any cannabis use in the last 30 days. Past 30-day cannabis use was assessed by timeline followback methods. Population: Due to technical issues with the timeline followback application, data was lost for 5 participants.
  Participants
    number analyzed (Participants) | 86 | 87 | 83 | 256
    (all) | 61 | 64 | 62 | 187
Cannabis: Median number of days used per week in last 30 days [Median (Inter-Quartile Range); unit: days per week] — The median number of days per week in which a participant used cannabis in the last 30 days. Cannabis use was assessed using timeline followback methods. Population: Due to technical issues with the timeline followback application, data was lost for 7 participants.
  days per week
    number analyzed (Participants) | 85 | 86 | 83 | 254
    (all) | 0.9 [0 to 4.3] | 2.1 [0 to 5.1] | 1.2 [0 to 4.8] | 1.4 [0 to 4.9]
Cannabis Use Disorders Identification Test- Revised (CUDIT-R) [Median (Inter-Quartile Range); unit: score on a scale] — The Cannabis Use Disorders Identification Test-Revised (CUDIT-R) is a screening designed to assess problematic cannabis use. It consists of 8 self-report items that measure frequency of use, symptoms of dependence, and the negative impacts of cannabis on daily life over the past six months. Each item is scored on a scale from 0 to 4, with higher scores indiciating greater severity of cannabis-related problems. The total score can range from 0 to 32, and a score of 8 or more suggests a potential cannabis use disorder. Population: A total score could not be calculated for two participants due to missing items.
  score on a scale
    number analyzed (Participants) | 87 | 87 | 85 | 259
    (all) | 6 [2 to 11.5] | 8 [3 to 14] | 8 [3 to 14] | 7 [3 to 13]
Alcohol: Past 30-day use [Count of Participants; unit: Participants] — Count of participants reporting any alcohol use in the last 30 days. Past 30-day alcohol use was assessed using timeline followback methods.
  Participants | 87 | 79 | 82 | 248
Alcohol: Median number of days used per week in last 30 days [Median (Inter-Quartile Range); unit: days per week] — The median number of days per week in which a participant used alcohol in the last 30 days. Past 30-day alcohol use was assessed using timeline followback methods. Population: Due to technical issues with the timeline followback application, data was lost for 12 participants.
  days per week
    number analyzed (Participants) | 83 | 85 | 81 | 249
    (all) | 1.4 [0.7 to 2.0] | 1.2 [0.5 to 1.9] | 0.9 [0.5 to 1.9] | 1.2 [0.5 to 1.9]
Alcohol Use Disorders Identification Test (AUDIT) [Median (Inter-Quartile Range); unit: score on a scale] — The Alcohol Use Disorders Identification Test (AUDIT) is a 10-item screening tool to assess problematic alcohol use. Scores range from 0 to 40, with higher scores indicating greater likelihood that alcohol use is negatively impacting health. Scores of 8-14 indicate likely harmful/hazardous drinking and scores of 15 or greater indicate a likely alcohol use disorder. Population: A total score could not be calculated for 4 participants due to missing items.
  score on a scale
    number analyzed (Participants) | 86 | 86 | 85 | 257
    (all) | 5 [3 to 9] | 7 [4 to 9] | 6 [4 to 10] | 6 [4 to 9]
Any self-reported psychiatric diagnosis [Count of Participants; unit: Participants] — Count of participants who self-reported any current psychiatric diagnosis. Self-reported psychiatric diagnoses were assessed via self-reported medical and psychiatric history.
  Participants | 60 | 61 | 55 | 176
Current Psychotropic Medication Use [Count of Participants; unit: Participants] — Count of participants who reported any current psychotropic medication use. Participants were asked to self-report all concomitant medications at each study visit.
  Participants | 33 | 33 | 33 | 99
Mood and Anxiety Symptoms Questionnaire (MASQ-D30) Total Score [Mean (Standard Deviation); unit: score on a scale] — Mood and Anxiety Symptoms Questionnaire (MASQ-D30) is a 30-item adaptation of the original 96-item MASQ, which instructs participants to rate how often in the past week they have experienced symptoms of depression and anxiety on a 5-point Likert scale from 1 ("not at all") to 5 ("extremely"). Total scores range from 30-150. Positive affect items are reverse-scored, and then a sum is calculated to reflect overall degree of mood and anxiety symptoms, with higher scores indicating more mood and anxiety symptoms.
  score on a scale | 57.8 (14.5) | 58.3 (14.8) | 58.6 (15.3) | 58.2 (14.8)
Mood and Anxiety Symptoms Questionnaire (MASQ-D30): General Distress Score [Mean (Standard Deviation); unit: score on a scale] — Mood and Anxiety Symptoms Questionnaire (MASQ-D30) is a 30-item adaptation of the original 96-item MASQ, which instructs participants to rate how often in the past week they have experienced symptoms of depression and anxiety on a 5-point Likert scale from 1 ("not at all") to 5 ("extremely"). The general distress subscale is calculated using 10 items and has a range of 10-50. Items are summed to calculate a total score. Higher scores represent greater distress from anxiety and depression symptoms.
  score on a scale | 17.4 (6.7) | 17.5 (6.0) | 18.8 (7.9) | 17.9 (6.9)

OUTCOME MEASURES:

1. Primary Outcome: Continuous 4-week Nicotine Vaping Abstinence at End of Treatment (Weeks 9-12)
Description: Point-prevalence abstinence from e-cigarette use was defined as self-report of no e-cigarette use since the last visit, bioverified by saliva cotinine <30 ng/ml. Continuous abstinence is defined as observed point-prevalence abstinence over specified study visits at weeks 9, 10, 11 and 12. Visits with self-reported abstinence missing bioverification were treated as missing, with missingness addressed via multiple imputation.
Time Frame: Assessments at study weeks 9, 10, 11, and 12
Measure: Count of Participants; unit: Participants
Arm/Group | Double Blind Varenicline (V+BC) | Double Blind Placebo (P+BC) | Single Blind Enhanced Usual Care (EUC)
Number analyzed (Participants) | 88 | 87 | 86
Participants | 45 | 12 | 5
Statistical Analysis 1: Comparison: Double Blind Varenicline (V+BC) vs Double Blind Placebo (P+BC); Test type: Superiority; p < 0.001, Regression, Logistic; Model fit to data from varenicline and placebo groups only, adjusted for sex and baseline E-cigarette Dependence Inventory score; Odds Ratio (OR) = 6.5, 95% CI 2-sided [3.0 to 14.1] — Adjusted odds ratio comparing varenicline (numerator) versus placebo (denominator)
Statistical Analysis 2: Comparison: Double Blind Varenicline (V+BC) vs Double Blind Placebo (P+BC) vs Single Blind Enhanced Usual Care (EUC); Test type: Superiority; p < 0.001, Regression, Logistic — The p-value is adjusted for multiple comparisons using per Benjamini & Hochberg (1995) across the primary outcome measure. Effects were deemed significant for p<0.05; Omnibus tests for any difference in abstinence rates across study groups, based on χ² Wald statistic and adjusted for sex and baseline ECDI score

2. Secondary Outcome: Seven-Day Point-Prevalence Nicotine Vaping Abstinence at End of Treatment (Week 12)
Description: Point-prevalence abstinence from e-cigarette use was defined as self-report of no e-cigarette use since the last visit, bioverified by saliva cotinine <30 ng/ml. Visits with self-reported abstinence missing bioverification were treated as missing, with missingness addressed via multiple imputation.
Time Frame: Study week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Double Blind Varenicline (V+BC) | Double Blind Placebo (P+BC) | Single Blind Enhanced Usual Care (EUC)
Number analyzed (Participants) | 88 | 87 | 86
Participants | 60 | 22 | 13
Statistical Analysis 1: Comparison: Double Blind Varenicline (V+BC) vs Double Blind Placebo (P+BC); Test type: Superiority; p < 0.001, Regression, Logistic — Benjamini-Hochberg multiplicity correction applied to p-values reported across family of five secondary analysis results (Varenicline vs Placebo comparisons of secondary abstinence outcomes, and omnibus tests of all three abstinence outcomes); [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 6.1, 95% CI 2-sided [3.1 to 12.3] — Adjusted odds ratio comparing varenicline (numerator) versus placebo (denominator)
Statistical Analysis 2: Comparison: Double Blind Varenicline (V+BC) vs Double Blind Placebo (P+BC) vs Single Blind Enhanced Usual Care (EUC); Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 2]

3. Secondary Outcome: Continuous Nicotine Vaping Abstinence Over Study Weeks 9 to 24
Description: Point-prevalence abstinence from e-cigarette use was defined as self-report of no e-cigarette use since the last visit, bioverified by saliva cotinine <30 ng/ml. Continuous abstinence defined as observed point-prevalence abstinence over specified study visits at weeks 9, 10, 11, 12, 16, 20, and 24. Visits with self-reported abstinence missing bioverification were treated as missing, with missingness addressed via multiple imputation.
Time Frame: Study weeks 9, 10, 11, 12, 16, 20, 24
Measure: Count of Participants; unit: Participants
Arm/Group | Double Blind Varenicline (V+BC) | Double Blind Placebo (P+BC) | Single Blind Enhanced Usual Care (EUC)
Number analyzed (Participants) | 88 | 87 | 86
Participants | 25 | 6 | 3
Statistical Analysis 1: Comparison: Double Blind Varenicline (V+BC) vs Double Blind Placebo (P+BC); Test type: Superiority; p = 0.001, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 6.0, 95% CI 2-sided [2.1 to 16.9] — Adjusted odds ratio comparing varenicline (numerator) versus placebo (denominator)
Statistical Analysis 2: Comparison: Double Blind Varenicline (V+BC) vs Double Blind Placebo (P+BC) vs Single Blind Enhanced Usual Care (EUC); Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 2]

4. Secondary Outcome: Minnesota Nicotine Withdrawal Scale (MNWS) Total Score (Weeks 1-12)
Description: Minnesota Nicotine Withdrawal Scale (MNWS) total scores over study weeks 1 to 12. The MNWS is an 8-item measure assessing the severity of nicotine withdrawal symptoms. Items are scored on an ordinal scale from 0 ("not at all") to 4 ("extreme") with total scores ranging from 0 to 32. Higher scores indicate greater severity of nicotine withdrawal symptoms. Missingness due to missed visits and/or dropout was addressed via multiple imputation.
Time Frame: Study weeks 1-12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Double Blind Varenicline (V+BC) | Double Blind Placebo (P+BC) | Single Blind Enhanced Usual Care (EUC)
Number analyzed (Participants) | 88 | 87 | 86
score on a scale
  Week 1 | 8.7 (6.2) | 10.6 (5.8) | 10.4 (5.8)
  Week 2 | 9.2 (6.3) | 10.6 (6.0) | 10.0 (5.9)
  Week 3 | 8.2 (6.4) | 10.5 (5.8) | 9.5 (5.8)
  Week 4 | 7.2 (5.7) | 10.9 (6.2) | 9.3 (5.6)
  Week 5 | 7.1 (6.0) | 9.2 (6.3) | 8.8 (5.9)
  Week 6 | 6.8 (6.0) | 8.2 (5.8) | 8.1 (6.0)
  Week 7 | 6.3 (6.0) | 8.5 (5.8) | 7.7 (5.3)
  Week 8 | 6.2 (5.6) | 7.9 (5.8) | 7.3 (5.8)
  Week 9 | 5.4 (5.0) | 7.6 (5.5) | 8.1 (6.1)
  Week 10 | 5.1 (5.2) | 6.8 (5.3) | 7.9 (5.9)
  Week 11 | 4.6 (5.0) | 6.6 (5.2) | 7.7 (5.5)
  Week 12 | 4.5 (4.5) | 7.0 (6.4) | 7.6 (5.5)
Statistical Analysis 1: Comparison: Double Blind Varenicline (V+BC) vs Double Blind Placebo (P+BC); Test type: Superiority; p = 0.001, Regression, Linear — Benjamini-Hochberg multiplicity correction applied to p-values reported across family of three secondary analysis results (Varenicline vs Placebo comparisons of secondary inventory outcomes); Models fit to data from varenicline and placebo groups only using GEE, adjusted for sex, baseline ECDI and outcome score, and quadratic trend of time; Mean Difference (Net) = -1.88, 95% CI 2-sided [-2.93 to -0.83] — Adjusted mean difference comparing varenicline versus placebo. Negative indicates larger mean in placebo
Statistical Analysis 2: Comparison: Double Blind Varenicline (V+BC) vs Double Blind Placebo (P+BC) vs Single Blind Enhanced Usual Care (EUC); Test type: Superiority; p < 0.001, Regression, Linear — [p-value comment as in outcome 4, analysis 1]; Models fit using GEE, adjusted for sex, baseline ECDI and outcome score, and quadratic time. Omnibus Wald test of any difference across study group

5. Secondary Outcome: Questionnaire of Vaping Craving (QVC) Total Scores (Weeks 1-12)
Description: Summed scores from the Questionnaire of Vaping Craving (QVC) over Study Weeks 1 to 12. The QVC is a 10-item self-rated validated measure (ranging from 10 to 70) of vaping craving that examines desire and intent to vape and anticipation of positive outcomes related to e-cigarette use, with higher scores indicating greater cravings to vape. Missingness due to missed visits and/or dropout are addressed with multiple imputation.
Time Frame: Study weeks 1-12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Double Blind Varenicline (V+BC) | Double Blind Placebo (P+BC) | Single Blind Enhanced Usual Care (EUC)
Number analyzed (Participants) | 88 | 87 | 86
score on a scale
  Week 1 | 34.1 (12.1) | 39 (12.2) | 37 (13)
  Week 2 | 29 (12.2) | 37.3 (13) | 36.6 (12.8)
  Week 3 | 25.8 (12.9) | 34.8 (12.1) | 34.1 (12.3)
  Week 4 | 22.8 (11.4) | 33.2 (13.4) | 34.1 (13.4)
  Week 5 | 20.4 (10.1) | 32.2 (12.8) | 32 (13.8)
  Week 6 | 19.3 (10.5) | 29.2 (13.1) | 32.5 (14)
  Week 7 | 18.9 (10.3) | 27.8 (14) | 31.2 (14.4)
  Week 8 | 17.8 (9.8) | 26.9 (13.6) | 30 (14.8)
  Week 9 | 17.1 (9.7) | 25.4 (13.1) | 31.2 (13)
  Week 10 | 15.9 (8.7) | 24 (12.2) | 30.4 (13.3)
  Week 11 | 16 (8.7) | 22.1 (11.5) | 28.9 (14.1)
  Week 12 | 14.4 (6.9) | 22 (11.2) | 28.1 (13.3)
Statistical Analysis 1: Comparison: Double Blind Varenicline (V+BC) vs Double Blind Placebo (P+BC); Test type: Superiority; p < 0.001, Regression, Linear — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 4, analysis 1]; Mean Difference (Net) = -6.76, 95% CI 2-sided [-9.08 to -4.45] — Adjusted mean difference comparing varenicline versus placebo. Negative indicates larger mean in placebo
Statistical Analysis 2: Comparison: Double Blind Varenicline (V+BC) vs Double Blind Placebo (P+BC) vs Single Blind Enhanced Usual Care (EUC); Test type: Superiority; p < 0.001, Regression, Linear — Benjamini-Hochberg multiplicity correction applied to p-values reported across family of three secondary analysis results (Omnibus tests of secondary inventory outcomes); Models fit using GEE, adjusted for sex, baseline ECDI and outcome score, and quadratic time. Omnibus Wald test of any difference across study groups

6. Secondary Outcome: Mood and Anxiety Symptoms Questionnaire (MASQ-D30) General Distress Subscore (Weeks 4, 8, and 12)
Description: Summed scores from the General Distress Subscale of the 30-Item Mood and Anxiety Symptoms Questionnaire (MASQ-D30) over Study Weeks 4,8, and 12. The General Distress subscale of the MASQ-D30 is a 10-item self-rated validated measure (ranging from 10 to 50) of non-specific symptoms of general distress or negative affect, with higher scores indicating a greater degree of general distress. Missingness due to missed visits and/or dropout was addressed with multiple imputation.
Time Frame: Study weeks 4, 8, 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Double Blind Varenicline (V+BC) | Double Blind Placebo (P+BC) | Single Blind Enhanced Usual Care (EUC)
Number analyzed (Participants) | 88 | 87 | 86
score on a scale
  Week 4 | 15.8 (5.8) | 19 (6.5) | 17.9 (6.6)
  Week 8 | 15.6 (6.3) | 16.9 (6.2) | 16.9 (6.2)
  Week 12 | 15.2 (5.8) | 16.6 (6.3) | 17 (6.9)
Statistical Analysis 1: Comparison: Double Blind Varenicline (V+BC) vs Double Blind Placebo (P+BC); Test type: Superiority; p = 0.008, Regression, Linear — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 4, analysis 1]; Mean Difference (Net) = -1.78, 95% CI 2-sided [-3.08 to -0.48] — Adjusted mean difference comparing varenicline versus placebo. Negative indicates larger mean in placebo
Statistical Analysis 2: Comparison: Double Blind Varenicline (V+BC) vs Double Blind Placebo (P+BC) vs Single Blind Enhanced Usual Care (EUC); Test type: Superiority; p = 0.02, Regression, Linear — Benjamini-Hochberg multiplicity correction applied to p-values reported across family of three secondary analysis results (Omnibus Wald test of secondary inventory outcomes); [statistical method as in outcome 5, analysis 2]

7. Secondary Outcome: Neuropsychiatric Adverse Event Inventory (NAEI) Elicited Adverse Events by Week 12
Description: The Neuropsychiatric Adverse Event Inventory (NAEI) is a structured interview used to assess neuropsychiatric adverse events. This outcome reports on the number of participants who reported at least one adverse event on the NAEI between the first study week (Week 1) to the end of treatment (Week 12).
Time Frame: Study weeks 1-12
Population: Analysis limited to participants who received randomized treatment. Because one participant randomized to placebo (P+BC) did not receive treatment, the denominator for the analysis is 86.
Measure: Count of Participants; unit: Participants
Arm/Group | Double Blind Varenicline (V+BC) | Double Blind Placebo (P+BC) | Single Blind Enhanced Usual Care (EUC)
Number analyzed (Participants) | 88 | 86 | 86
Participants | 71 | 61 | 78
Statistical Analysis 1: Comparison: Double Blind Varenicline (V+BC) vs Double Blind Placebo (P+BC); Test type: Superiority; p = 0.16, Fisher Exact
Statistical Analysis 2: Comparison: Double Blind Varenicline (V+BC) vs Single Blind Enhanced Usual Care (EUC); Test type: Superiority; p = 0.083, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 24 weeks.
Description: Analysis limited to participants who received randomized treatment. Because one participant randomized to placebo (P+BC) did not receive treatment, the denominator for the analysis is 86.
Arm/Group | Double Blind Varenicline (V+BC) | Double Blind Placebo (P+BC) | Single Blind Enhanced Usual Care (EUC)
All-Cause Mortality (participants affected / at risk) | 0/88 | 0/86 | 0/86
Serious Adverse Events (participants affected / at risk) | 1/88 | 3/86 | 1/86
Other Adverse Events (participants affected / at risk) | 78/88 | 73/86 | 69/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double Blind Varenicline (V+BC) (N=88) | Double Blind Placebo (P+BC) (N=86) | Single Blind Enhanced Usual Care (EUC) (N=86)
Psychiatric Hospitalization (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1)
Motor Vehicle Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Snowboarding Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double Blind Varenicline (V+BC) (N=88) | Double Blind Placebo (P+BC) (N=86) | Single Blind Enhanced Usual Care (EUC) (N=86)
Cold symptoms (Respiratory, thoracic and mediastinal disorders) | 42 (69) | 29 (36) | 36 (53)
Nausea and vomiting symptoms (Gastrointestinal disorders) | 51 (82) | 23 (29) | 5 (6)
Vivid dreams (Psychiatric disorders) | 34 (46) | 14 (16) | 0 (0)
Insomnia (Nervous system disorders) | 27 (38) | 16 (21) | 8 (9)
Bloating (Gastrointestinal disorders) | 28 (32) | 22 (26) | 2 (2)
Anxiety disorders and symptoms (Psychiatric disorders) | 22 (37) | 28 (51) | 32 (49)
Mood disorders and disturbances (Psychiatric disorders) | 22 (32) | 28 (35) | 22 (31)
Constipation (Gastrointestinal disorders) | 14 (17) | 9 (10) | 3 (3)
Headache (Nervous system disorders) | 14 (16) | 19 (20) | 7 (8)
Withdrawal symptom (General disorders) | 7 (7) | 7 (7) | 8 (11)
Appetite increased (General disorders) | 5 (5) | 3 (3) | 6 (6)
Chest pain (General disorders) | 0 (0) | 1 (1) | 5 (5)

LIMITATIONS AND CAVEATS:
The sample size was underpowered to detect the observed difference in the exploratory comparison between P+ BC and EUC. Results may not generalize to those who regularly use both combustible tobacco and vaped nicotine.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2024-01-10): https://cdn.clinicaltrials.gov/large-docs/92/NCT05367492/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-13): https://cdn.clinicaltrials.gov/large-docs/92/NCT05367492/SAP_001.pdf
  • Informed Consent Form (2024-10-09): https://cdn.clinicaltrials.gov/large-docs/92/NCT05367492/ICF_002.pdf